CLINICAL TRIAL: NCT03102814
Title: The BRIDGE Trial: A Multicenter RCT to Improve Continuity and Quality in Rehabilitation of People With Rheumatic and Musculoskeletal Diseases
Brief Title: The BRIDGE Rehabilitation Trial
Acronym: BRIDGE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Resource Center for Rehabilitation in Rheumatology (Other)
Collaborators: Sørlandet Hospital (Unknown); Vikersund Rehabilitation Centre (Unknown); Muritunet Rehabilitation Centre (Unknown); Valnesfjord Rehabilitation Centre (Unknown); Meråker Rehabilitation Centre (Unknown); Rehab Vest Rehabilitation Centre (Unknown); Lillehammer Rheumatism Hospital (Unknown); Haugesund Rheumatism Hospital (Other)
Responsible Party: Principal Investigator, Ingvild Kjeken, Professor, National Resource Center for Rehabilitation in Rheumatology
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: Project nr 97033
Record Dates: First submitted 2017-03-31; First posted 2017-04-06 (Actual); Last update posted 2020-03-02 (Actual); Status verified 2020-02

CONDITIONS: Musculoskeletal Disease
MeSH Terms: conditions — Musculoskeletal Diseases

STUDY DESIGN:
Intervention Model Description: In order to evaluate the effects of the BRIDGE program, a stepped wedge cluster randomized controlled trial will be conducted. In the trial, participating centres switch from control (current rehabilitation program) to intervention phase (adding the BRIDGE program to the current program) in a randomized order. All centres start the trial simultaneously and act as controls until the point in time they are randomized to crossover from control to intervention, and all centres deliver the intervention by the end of inclusion.
  The stepped wedge design is suitable for a phased evaluation approach, where it is difficult to deliver two parallel interventions.
Who Masked: Investigator
Masking Description: Due to the nature of the study intervention, it is not possible to blind participants or the health care providers. However, the statistician who will perform the main statistical analyses will be blinded to group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Current rehabilitation program (Active Comparator): The control group will receive the rehabilitation program currently provided at each participating centre at the start of the study.
  Interventions: Behavioral: Current rehabilitation
- BRIDGE rehabilitation program (Experimental): In intervention phase, the BRIDGE program will be added to the current program.
  Interventions: Behavioral: The BRIDGE program

INTERVENTIONS:
Behavioral: Current rehabilitation — The control group will receive the rehabilitation currently offered at each of the participating centers.
  Arms: Current rehabilitation program
Behavioral: The BRIDGE program — The experimental group will additionally receive the BRIDGE program, which comprises motivational interviewing, structured goal-setting, tailored follow-up, plans for self-management, and individualised written feedback that participants can use to monitor their progress and share with important care givers.
  Arms: BRIDGE rehabilitation program

SUMMARY:
The main aim of this multi-centre stepped wedge randomized controlled trial is to improve the quality, professional practice and cost-effective utilization of health care resources by evaluating if a new rehabilitation program aimed at bridging gaps in rehabilitation across levels of care may increase and/or prolong the effect of rehabilitation.

DETAILED DESCRIPTION:
The goal of rehabilitation is to help people to reach and maintain their optimal functioning and coping capabilities, and to promote independence and participation in society. According to current political documents, there are large variation in the content and quality of rehabilitation in Norway, and systems to improve coordination and communication are needed.

This trial is a collaborative project between eight centres across Norway, investigating whether a new program aimed at bridging gaps in rehabilitation across levels of care increase and/or prolong the effect of rehabilitation for people with rheumatic and musculoskeletal diseases. Additionally, we will use a newly developed set of quality indicators to monitor and compare the quality of rehabilitation across different centres, and explore relationships between adherence to structure and process indicators and the outcomes of rehabilitation.

The effects will be evaluated in a multi-centre stepped wedge randomized controlled trial, where participating centres switch from control (current rehabilitation program) to intervention phase (adding the BRIDGE program to the current program) in a randomized order. Primary outcome is goal attainment after seven months, and secondary outcomes are health related quality of life and function.

The results will give insight in the content and organisation of current rehabilitation programs, what follow-up people want and receive in primary care, their planned and completed efforts to implement and maintain life style changes, and predictors for improvement following rehabilitation in specialist health care. Results will also have consequences on how rehabilitation is to be organized in the future regarding follow-up and coordination across levels of care.

The study has been developed in close collaboration with patient research partners, clinicians and international experts, who will also contribute in the process of integrating study results in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* inflammatory rheumatic disease or osteoarthritis or fibromyalgia or low back pain or wide spread pain or osteoporosis. Having a good understanding of Norwegian and having a bank-ID

Exclusion Criteria:

* Cognitive impairment or severe psychiatric disorder

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 381 (Actual)
Dates: Start 2017-08-15 (Actual); Primary Completion 2019-08-30 (Actual); Study Completion 2019-08-30 (Actual)

PRIMARY OUTCOMES:
Goal attainment measured by the Patient Specific Functional Scale | One year
  Goal attainment will be measured by the Patient Specific Functional Scale

SECONDARY OUTCOMES:
Health-related quality of life measured by the EQ5D | One year
  Health-related quality of life will be measured by the EQ5D
Physical function measured by the 30 sec sit to stand test | One year
  Physical function will be measured by the 30 sec sit to stand test

OTHER OUTCOMES:
Pain measured on a numeric rating scale | One year
  Pain will be measured on a numeric rating scale
Fatigue measured on a numeric rating scale | One Year
  Fatigue will be measured on a numeric rating scale
Motivation for goal attainment measured on a numeric rating scale | Baseline
  Motivation for goal attainment will be measured on a numeric rating scale
Function in daily activities measured by the Hannover Functional Ability Questionnaire | One year
  Daily activities will be measured by the Hannover Functional Ability Questionnaire
Coping measured by the Effective Musculoskeletal Consumer Scale | One year
  Coping will be measured by the Effective Musculoskeletal Consumer Scale
Mental health measured by the Hopkins Symptom Checklist | One year
  Mental health will be measured by the Hopkins Symptom Checklist
Participation measured by participation scale in COOP/WONCA | One year
  Participation will be measured by participation scale in COOP/WONCA

CONTACTS AND LOCATIONS:
Overall Officials: Tore K Kvien, PhD, Study Director — Diakonhjemmet Hospital
Locations (8):
- Norway (8):
  - Valnesfjord Rehabilitation Centre, Valnesfjord, Valnesfjord
  - Sørlandet Hospital, Arendal
  - Haugesund Rheumatism Hospital, Haugesund
  - Rehabilitering Vest, Haugesund
  - Lillehammer Rheumatism Hospital, Lillehammer
  - Meråker rehabilitation centre, Meråker
  - Muritunet Rehabilitation Centre, Valldal
  - Vikersund Rehabilitation Centre, Vikersund

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sand-Svartrud AL, Berdal G, Azimi M, Bo I, Dager TN, Eppeland SG, Fredheim GO, Hagland AS, Klokkeide A, Linge AD, Sexton J, Tennebo K, Valaas HL, Mjosund K, Dagfinrud H, Kjeken I. Associations between quality of health care and clinical outcomes in patients with rheumatic and musculoskeletal diseases: a rehabilitation cohort study. BMC Musculoskelet Disord. 2022 Apr 15;23(1):357. doi: 10.1186/s12891-022-05271-3. PMID 35428256
- [Derived] Sand-Svartrud AL, Berdal G, Azimi M, Bo I, Dager TN, Eppeland SG, Fredheim GO, Hagland AS, Klokkeide A, Linge AD, Tennebo K, Valaas HL, Aasvold AM, Dagfinrud H, Kjeken I. A quality indicator set for rehabilitation services for people with rheumatic and musculoskeletal diseases demonstrates adequate responsiveness in a pre-post evaluation. BMC Health Serv Res. 2021 Feb 20;21(1):164. doi: 10.1186/s12913-021-06164-2. PMID 33610174